CLINICAL TRIAL: NCT04512508
Title: Anal Injury Screening for High Risk HPV in Population With Susceptibility to Anal Cancer Development
Brief Title: Anal Injury Screening for High Risk HPV
Acronym: AnalTest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Principal Investigator, Dr. Carlos E. Aranda Flores, Surgeon, specialty in oncology, Hospital General de México Dr. Eduardo Liceaga
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DI/20/111/03/11
Record Dates: First submitted 2020-07-30; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Anal Injury; Anal Cancer
Keywords: Anal cancer; Anal test; Anoscopy; HPV
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomized and consecutive number will be assigned. If it is a non-number, the self-test will be performed first, followed by liquid cytology and then anoscopy. If it is a even number, first the liquid cytology will be performed, then the autotoma and the anoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1, HIV negative patients. (Other): Only HIV negative patients
  Interventions: Diagnostic Test: Self test sample
- Group 2, HIV positive patients (Other): Only HIV positive patients
  Interventions: Diagnostic Test: Self test sample

INTERVENTIONS:
Diagnostic Test: Self test sample — Self test sample, DNA analysis, Biopsy and Anoscopy
  Other Names: Citology sample

SUMMARY:
The diagnosis of anal cancer is superior with the Anal Test system compared to liquid cytology and anoscopy.

DETAILED DESCRIPTION:
DESIGN METHODOLOGY: Prospective, cross-sectional, comparative, double-blind, randomized.

STUDY POPULATION:

Group 1, 250 HIV negative patients (150 men and 100 women) from the oncology service who agree to participate in the study and with a negative diagnosis for HIV made at the Infectious Diseases Service.

Group 2, 250 HIV positive patients (150 men and 100 women) attended by the Infectious Disease Service diagnosed with HIV positive. The sample size was adjusted to the donation of 500 Anal Test devices and the subsequent molecular determinations for each sample.

PROCEDURE:

In this study, men and women between 30 and 65 years old with active sexual life and who are susceptible to the development of anal cancer can participate.

1. Immunosuppressed patients, a) infected with the human immunodeficiency virus, HIV or b) by medication after receiving an organ transplant.
2. Individuals who have or have had anal intercourse. Women with a history of cervical, vulva, or vaginal cancer.

PLANNED ACTIVITIES:

First: Candidate patients who meet the inclusion criteria will have an explanation of the importance of their participation in this protocol, all their doubts will be resolved and they will be asked to sign the letter of informed consent with witnesses.

Second: After signing the letter of consent, the service provider will make a questionnaire to know the clinical characteristics and identification of the patient, they will be assigned a consecutive number.

If assignation is a non-number, the self-test will be performed as the first in sequence, followed by liquid cytology and then anoscopy.

If assignation is an even number, the liquid cytology will be done as the first in sequence, followed by self-test and the anoscopy.

* For the Self-Test: the patient will be given the Anal Test medical device with the following recommendations: a) washing of patient hands, b) removing the plastic packaging from the device, c) removing the cover, d) Holding it by the handle, the device will be inserted into the anus, e) patient will be left intro-anal for 30 seconds and then it will be rotated 180 degrees, f) it will slowly withdraw the device and g) it will be delivered to the assistant nurse.
* The nurse will put the device (with the sample) in a tube with 5 ml of PreservCyt solution and close it tightly.
* The tube with the device and the sample will be kept at room temperature until transport to the laboratory for processing and obtaining results.
* The patient will answer a satisfaction questionnaire.
* An appointment will be given three weeks later to grant the result.

Third:

Processing of samples and issuance of results will be done in an external laboratory outside the Hospital General de México. In the Molecular Biology Laboratory, the coded samples will be processed as follows:

1. DNA will be extracted using the Abbott Real-Time Polymerase Chain Reaction (RT-PCR) technology procedures, with the m2000 system. Presence and identification will be determined for HPV-Ar 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
2. Only the positive samples from the first step; mRNA will be extracted and the viral oncology proteins expression of the E6 and E7 will be quantified for the following specific HPV-Ar 16, 18, 31, 33, 45, 52 and 58 by Real-Time Polymerase Chain Reaction (RT-PCR). The results of the laboratory studies will be sent to the responsible investigator.
3. Processing of samples in an external laboratory outside the Hospital General de México and issuance of results. In the Molecular Biology Laboratory, the coded samples will be processed as follows:

   1. DNA will be extracted using the Abbott Real-Time Polymerase Chain Reaction (RT-PCR) technology procedures, with the m2000 system. The presence and identification will be determined for HPV-Ar 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
   2. Only the positive samples from the first step; mRNA will be extracted and the expression of the viral oncology proteins E6 and E7 will be quantified for the following specific HPV-Ar 16, 18, 31, 33, 45, 52 and 58 by Real-Time Polymerase Chain Reaction (RT-PCR). The results of the laboratory studies will be sent to the responsible investigator.

Fourth:

If they are positive to HPV-Ar, investigator will follow-up patient to corroborate the elimination or persistence of the HPV infection (surveillance). Patients who are positive for E6 and E7 messenger ribonucleic acid (mRNA) will be cited for high-resolution anoscopy and biopsy, negative patients will be under surveillance. Patients who are normal or with Low grade Intraepithelial Lesion (lSIL) (NIA1) by cytology will be under surveillance. High grade Intraepithelial Lesion (HSIL) patients (NIA2 and NIA3) will be scheduled for high-resolution anoscopy and biopsy.

STATISTICAL ANALYSIS Statistical results will be reported first in a descriptive way, reporting means and standard deviations of the main study variables, as well as percentages of the presence of high-risk human papillomavirus analyzed in this investigation. Bi-variate comparative tests such as t-Student or Chi-square tests will be applied to identify possible differences between the group of people with the presence/absence of high-risk viruses and demographics and clinical variables such as the presence of HIV. When there is no normality, the non-parametric Mann-Whitney U test will be applied. Linear correlations will be analyzed with the Spearman and Pearson correlation tests depending on the type of analyzed variables. Data concordance analysis such as the kappa test will be performed because due to presence of human papillovirus HPV-Ar sub-types as well as lesion type compared to the results of liquid anal cytology that in this study the investigators will consider our "gold standard", in addition to perform sensitivity, specificity, positive and negative predictive value tests. Finally, and although it is not part of our main objectives, the investigators will analyze the possible associate risk factors with the presence of high-risk human papillovirus (HPV) using logistic regression models.

ETHICAL ASPECTS AND BIOSECURITY. ETHICS. What is indicated in relation to ethics on human studies will be strictly followed according to Regulations of the General Law of Health in Matters of Health Research of Mexico, and the Declaration of Helsinki, considering subsequent versions.

INFORMED CONSENT LETTER. SAFETY The subject under study will have complete information on the procedures that will be carrying out. The studies will be done exclusively with the assistance of the authorized research team and in consulting rooms belonging to the Oncology Service. If the subject under study expresses his desire not to participate in the process, it will be suspended immediately.

All the studies to be carried out on the patient are totally safe and innocuous.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 30 and 65 years old.
* They agree to participate in the study and sign informed consent.
* They have not received previous treatments for HPV or had previous intraepithelial lesions or anal cancer.
* Immunosuppressed patients.
* Women with LIAG of the genital tract (cervix, vagina, or vulva).
* Patients who have had anal intercourse

Exclusion Criteria:

* Patients sexually inactive
* Subjects who had anal sex in less than 24 hours prior to the study.
* Patients with local medication application (enemas, suppositories).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-08-30 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of positive results for Anal Test system versus anal liquid cytology and anoscopy for the presence of high-risk human papillomaviruses | 12 months
  Statistical difference for percentages of the presence of high-risk human papillomaviruses between self-test versus liquid anal cytology.

SECONDARY OUTCOMES:
Number of predictive value for positive and negative results for self-test versus liquid cytology results | 12 months
  Statistical difference To compare predictive positive and negative value by self-test versus liquid anal cytology.
Number and percentage of patients with anal intraepithelial lesions caused by HPV-Ar infection compared between HIV-positive and HIV-negative patients | 12 months
  Difference for anal intraepithelial lesions caused by HPV-Ar infection between HIV-positive and HIV-negative patients
Number and percentage of LSIL and HSIL for patients using self-test (by presence of mRNA for viral proteins E6 and E7) compared to number and percentage of LSIL and HSIL for patients with liquid cytology or with results by biopsy. | 12 months
  Number and frequency of LSIL and HSIL concordant between self-test and by liquid cytology and anoscopy or with biopsy results in positive patients for viral DNA.
Number and percentage of patients to have a positive opinion to use Self-Test system. | 12 months
  A survey will be applied to assess Anal Tests system acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Luis G Molina Fernández de Lara, Study Chair — Hospital General de México Eduardo Liceaga
Locations (1):
- Hospital General de México Eduardo Liceaga, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No